CLINICAL TRIAL: NCT06056869
Title: Effect of Hyoscine- Bromide on Duration of the First Stage of Labor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS 503/2023
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Labor
MeSH Terms: interventions — Butylscopolammonium Bromide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- buscopan group (Active Comparator): will receive 2 ml (40 mg) of hyoscine butylbromide
  Interventions: Drug: hyoscine butylbromide
- control group (Placebo Comparator): will receive 2 ml of normal saline
  Interventions: Other: normal saline

INTERVENTIONS:
Drug: hyoscine butylbromide — will be given during first stage of labor intravenously
  Arms: buscopan group
Other: normal saline — placebo
  Arms: control group

SUMMARY:
Spasmolytic drugs are frequently used in delivery rooms to overcome cervical spasms and thus reduce the duration of labor. The aim of this randomized double blind placebo controlled trial is to study the efficacy of hyoscine butylbromide (HBB) for shortening of the first stage of labor in primigravid women.

ELIGIBILITY:
Inclusion Criteria:

1. Primigravid women.
2. Singleton pregnancy.
3. Presenting by the vertex.
4. Gestational age between 37 and 42 weeks
5. In active phase of labor with a cervical dilatation between 4-5 cm, with either intact membranes or spontaneous rupture of membranes for less than 12 h

Exclusion Criteria:

1. Previous uterine scarring.
2. Malpresentation.
3. Antepartum hemorrhage.
4. Labor induction
5. Contraindication to vaginal delivery.
6. Contraindication to hyoscine.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
duration of first stage of labor | 6 months
  duration

CONTACTS AND LOCATIONS:
Overall Officials: Maii Nawara, Principal Investigator — Associate professor
Locations (1):
- Ain Shams University maternity hospital, Cairo, Cairo/القاهرة, Egypt

IPD SHARING:
Plan to Share IPD: Yes
will be available with principal investigator if required